CLINICAL TRIAL: NCT00494286
Title: Treatment of Child Physical Abuse: An Effectiveness Trial (PFF)
Brief Title: Abuse-Focused Cognitive Behavioral Therapy for Children Who Have Been Physically Abused
Acronym: PFF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Kolko, Professor of Psychiatry, Psychology, and Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH074737 (NIH); R01MH074737 (NIH); DSIR CT-C
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Child Abuse
Keywords: Abuse Focused Cognitive Behavioral Therapy; Treatment Effectiveness Research; Treatment Dissemination
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AF-CBT (Experimental): Participants will receive abused-focused cognitive behavioral therapy
  Interventions: Behavioral: Abused-focused cognitive behavioral therapy (AF-CBT)
- TAU (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Abused-focused cognitive behavioral therapy (AF-CBT) — Practitioners will be randomly assigned to provide the AF-CBT treatment for 3 to 6 months. Patient participants will continue to see their regular practitioner, but will receive AF-CBT at treatment visits. Practitioners who are assigned to AF-CBT will first receive training in the treatment method. The training curriculum will include a published treatment book, intensive training sessions, which will occur weekly for 8 hours over 4 weeks, handouts that illustrate key therapeutic information and exercises, and ongoing case consultation reviews for 5 months.
  Arms: AF-CBT
Behavioral: Treatment as usual (TAU) — This condition consists of those practitioners in each agency who will not receive study training in AF-CBT. These practitioners will simply provide services as available within their agencies.
  Arms: TAU

SUMMARY:
This study will determine the effectiveness of abuse-focused cognitive behavioral therapy that is provided by a community health clinic in addressing the behavioral and emotional health needs of children and adolescents whose parents have used physical disciplinary action.

DETAILED DESCRIPTION:
Child physical abuse is a common public health problem that has been associated with significant psychosocial and physical health problems among children. Abuse-focused cognitive-behavioral therapy (AF-CBT) has been identified as an effective treatment strategy for dealing with child physical abuse. The main component of AF-CBT, cognitive behavioral therapy (CBT), is a type of psychotherapy in which everyday thoughts and behaviors are modified to improve mental health problems, such as depression or anxiety. AF-CBT uses CBT techniques to specifically focus on improving the mental health problems associated with physical abuse. In this study, AF-CBT will incorporate individual and family CBT and will be adapted by community practitioners to maximize its effectiveness in a community health care setting. This study will determine the effectiveness of AF-CBT, provided by a community health clinic, in addressing the behavioral and emotional health needs of children and adolescents whose parents have used physical disciplinary action.

Participants in this study will include practitioners, their supervisors, and their patients. Practitioners will be randomly assigned to provide either treatment as usual (TAU) or the AF-CBT intervention for 3 to 6 months. Patient participants will continue to see their regular practitioner, but will receive the type of treatment to which their practitioner has been assigned. Practitioners who are assigned to TAU will continue to attend training workshops or seminars as a part of their clinics' routine policies and their current personal practices. Practitioners who are assigned to AF-CBT will first receive training in the treatment method. The training curriculum will include a published treatment book, intensive training sessions, which will occur weekly for 8 hours over 4 weeks, handouts that illustrate key therapeutic information and exercises, and ongoing case consultation reviews for 5 months.

Parent and child participants will meet with practitioners at times to be decided based on individual patient needs. All parents and children will be asked to participate in interviews to assess symptoms and outcomes before attending any treatment sessions with the practitioner, 6 months, 12 months, 18 months,and 30 months after baseline. Parents and children will also complete questionnaires each time they meet with the practitioner. This study will also assess the ability of the practitioners and supervisors to carry out AF-CBT.

ELIGIBILITY:
Inclusion criteria:

* Child is between 5 and 15 years of age
* Any one of the following child discipline criteria are met within the past 12 months:

  1. the parent reports that the child has been the target of physical force/contact (e.g. discipline, punishment),
  2. the parent reports that the child has been the target of other acts that place the child at-risk for physical harm/injury (including threats of injury or harm) or
  3. an allegation or report of suspected physical abuse of this child was made to child welfare regardless of the outcome;
* Child and caregiver (preferably, not necessarily, the offending or at-risk caregiver, and regardless of whether they live together currently), will participate in services, and should be able to make progress in the proposed agency services;
* Parent/legal guardian must agree to informed consent for child and there is no immediate plan for a change in parental rights (e.g., child going to pre-adoptive foster care).

Exclusion Criteria:

* Child or parent is identified by agency staff as exhibiting serious psychological or intellectual impairment that would prevent minimal participation or progress in treatment (e.g., severe drug dependence, active psychosis, or pervasive developmental disorder)
* Child is in placement without access to a legal guardian who can provide informed consent OR a change in parental rights is likely to occur in the near future

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2006-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Family outcomes, including client engagement in service | Measured at baseline and Months 6, 12, 18, 24, and 30
Mental health functioning (symptom improvement, family support, more appropriate parenting practices) and outside service use (social service system contact or child placement/disruption) | Measured at baseline and Months 6, 12, 18, 24, and 30
Child welfare status (recidivism or re-injury rates) | Measured at baseline and Months 6, 12, 18, 24, and 30

SECONDARY OUTCOMES:
Practitioner knowledge about treatment | Measured at baseline and Months 6, 12, 18, 24, and 30
Practitioner competency and patient's satisfaction with treatment | Measured at baseline and Months 6, 12, 18, 24, and 30

CONTACTS AND LOCATIONS:
Overall Officials: David J. Kolko, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Bellefield Towers, Pittsburgh, Pennsylvania, United States